CLINICAL TRIAL: NCT02488083
Title: Clinical Study to Evaluate the Performance of the UltraShape Device for Thighs Fat and Circumference Reduction vs. Control
Brief Title: UltraShape Device for Thigh Fat and Circumference Reduction vs. Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF17991
Record Dates: First submitted 2015-05-26; First posted 2015-07-02 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Unwanted Thigh Fat
Keywords: non-invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all subjects treated by UltraShape (Experimental): all the patients undergo fat reduction treatment by UltraShape
  Interventions: Device: Ultrashape

INTERVENTIONS:
Device: Ultrashape — circumference reduction
  Other Names: fat reduction

SUMMARY:
UltraShape Device for Thigh Fat and Circumference Reduction: Prospective, blinded, one arm, baseline-controlled clinical study for the evaluation of the UltraShape treatment for non-invasive fat and circumference reduction.

DETAILED DESCRIPTION:
UltraShape Device for Thigh Fat and Circumference Reduction- Up to 60 healthy adult volunteers seeking for noninvasive thighs circumference reduction, male and females, 18 to 60 years of age from up to four investigational sites.

Eligible subjects will receive 3 bi-weekly treatments (2 weeks interval) on one randomized thigh with the UltraShape device according to the study protocol. The other thigh will not be treated during the main study phase (and serve as control).

The subjects will return for 3 follow up visits: four weeks (4wk FU), eight weeks (8wk FU) and 16 weeks (16wk FU) after the last treatment.

Total expected study duration: 20-22 weeks. Should the subject choose to receive additional optional treatments on the untreated side, up to three bi-weekly treatments will be performed upon study completion at no cost to the subject while changing total study duration to 24-26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Female and male subjects,18 and 60 years of age at the time of enrolment
3. Fitzpatrick Skin Type I to VI.
4. Fat thickness of at least 1.5 cm in the treated area (measured by calibrated caliper).
5. BMI interval: BMI in range of 22- 30 (normal to overweight, but not obese).
6. If female, not pregnant or lactating, must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
7. In addition, negative urine pregnancy test as tested before each treatment and at the last follow-up visit for women with child-bearing potential (e.g. not menopause).
8. General good health confirmed by medical history and skin examination of the treated area.
9. Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
10. Willingness to refrain from a change in diet/ exercise/medication regimen for the entire course of the study.
11. Willing to have photographs and images taken of the treated areas to be used, de-identified in evaluations, publications and presentations.

Exclusion Criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator, abdominal aortic aneurism
2. Known hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease
3. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions
4. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
5. Having a permanent implant in the treated area, such as metal plates or an injected chemical substance such as silicone
6. Having undergone any other surgery in the treated areas within 12 months of treatment or during the study, including liposuction
7. Previous body contouring procedures in the treatment area within 12 months
8. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing
9. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
10. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area
11. Very poor skin quality (i.e., severe laxity)
12. Abdominal wall diastasis or hernia on physical examination
13. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
14. Obesity (BMI bigger than 30)
15. Childbirth within the last 12 months or breastfeeding women. Any acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study
16. Unstable weight within the last 6 months (i.e tolerance of 3% weight change in the prior six months)
17. Inability to comply with circumference measurement procedure (e.g., inability to hold breath for the required duration).
18. Participation in another clinical study within the last 6 months.
19. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
evaluate the efficacy of the UltraShape device by evaluating the non-invasive fat and circumference reduction | 8 weeks up to 20 weeks

SECONDARY OUTCOMES:
safety issues assessed by The number, severity and type of any adverse event recorded throughout the study and post treatment (immediate and delayed response) | day 0 up to 20 weeks
thigh circumference reduction | four weeks (4wk FU), eight weeks (8wk FU) and 16 weeks (16wk FU) after the last treatment,
  significant thigh circumference reduction post UltraShape treatments. Reduction will be calculated at each follow-up visit (4wk FU, 8wk FU and 16wk FU) versus baseline and versus control thigh.
thigh fat thickness reduction by ultrasound | day 0, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 20 weeks
  fat thickness reduction post UltraShape treatments as measured by caliper and by Ultrasound device
thigh fat thickness reduction by caliper | day 0, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 20 weeks
  thigh fat thickness reduction
Subject satisfaction by questionnaire | 8 weeks, 12 weeks, 20 weeks
  Satisfaction assessment will be performed independently by the subject himself
Comfort level by NSR scale | day 0, 2 weeks, 4 weeks
  Comfort level during treatment will be performed post each treatment
Investigator satisfaction by questionnaire | 8 weeks, 12 weeks, 20 weeks
  assessment comparing before and after photos using the 5-Point Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Robert Weiss, MD, Principal Investigator — Maryland Laser Skin and Vein Institute
Locations (3):
- United States (3):
  - Coleman Center for Cosmetic Dermatologic Surgery, Metairie, Louisiana
  - Maryland Laser, Skin, & Vein Institute, Baltimore, Maryland
  - Skin Laser & Surgery Specialist of NY/NJ, Hackensack, New Jersey

REFERENCES:
- [Background] Ascher B. Safety and efficacy of UltraShape Contour I treatments to improve the appearance of body contours: multiple treatments in shorter intervals. Aesthet Surg J. 2010 Mar;30(2):217-24. doi: 10.1177/1090820X09360692. PMID 20442099
- [Background] Teitelbaum SA, Burns JL, Kubota J, Matsuda H, Otto MJ, Shirakabe Y, Suzuki Y, Brown SA. Noninvasive body contouring by focused ultrasound: safety and efficacy of the Contour I device in a multicenter, controlled, clinical study. Plast Reconstr Surg. 2007 Sep;120(3):779-789. doi: 10.1097/01.prs.0000270840.98133.c8. PMID 17700131